CLINICAL TRIAL: NCT03258580
Title: Sociocultural & Biobehavioral Influences on Pain Expression and Assessment
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: 170155; 17-AT-0155
Record Dates: First submitted 2017-08-22; First posted 2017-08-23 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-12-01

CONDITIONS: Normal Physiology; Healthy Volunteers; Pain
Keywords: Pain; Visual Analogue Pain Scale; Healthy Volunteer; EYE TRACKING; Eye Movement
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Substudy 1: All participants (Experimental): Measuring facial response to painful stimulation.
  Interventions: Device: Medoc thermal stimulator; Device: Electric shock stimulator; Device: Cold water bath
- Substudy 2: Healthy volunteers (No Intervention): Measuring pain assessment accuracy
- Substudy 3: Control (No Intervention): Subjects will judge stimuli with the same instructions as Sub-Study 2 (which provides a test of replication).
- Substudy 3: Feedback Group (Experimental): Participants in substudy 3's Feedback Group will be informed about their performance after every trial when making judgments about other people's pain.
  Interventions: Behavioral: Pain assessment performance feedback

INTERVENTIONS:
Device: Medoc thermal stimulator — Heat pain stimulation for substudy 1
  Arms: Substudy 1: All participants
Device: Electric shock stimulator — Electric pain stimulation for substudy 1
  Arms: Substudy 1: All participants
Device: Cold water bath — Cold pain stimulation for substudy 1
  Arms: Substudy 1: All participants
Behavioral: Pain assessment performance feedback — Participants in substudy 3's Feedback Group will be informed about their performance after every trial when making judgments about other people's pain.
  Arms: Substudy 3: Feedback Group

SUMMARY:
Objective

The current proposal investigates behavioral, psychophysiological, and social processes that may help explain biases and disparate outcomes in pain. Health disparities, or health outcomes that adversely affect disadvantaged populations, are pervasive and apparent in many diseases and symptoms, including pain. Pain is the number one reason individuals seek medical treatment. Health disparities in pain encompass both differences in pain experience and treatment for pain. For instance, research indicates that Black individuals report increased pain and have reduced pain tolerance relative to White individuals, yet doctors are less likely to treat minority patients pain and underestimate their pain experience. This project aims to address this systemic discrepancy by focusing on interpersonal processes that may contribute to these disparities, including socially-relevant responses to pain (i.e. pain expression) and pain assessment (e.g. visual attention). The proposed research aims to determine whether the study of pain expressions and their assessment can yield insights on how social factors shape pain and its treatment. Further, we test the efficacy of potential interventions designed to improve accuracy and reduce biases in pain assessment. If successful, this work will form the foundation of a new research program that will link the field of pain research with the field of social neuroscience, and forge new insights on the critical problem of health disparities in pain.

Study population

We will accrue up to 700 total healthy volunteers to target 240 completers

Design

Our overall aim is to understand how social factors influence the assessment and management of pain, and to gain insight into psychosocial processes that may underlie health disparities in pain. We propose a series of studies designed to test these links. First, we will measure pain perception and physiological responses to painful stimuli in a diverse group of individuals to test for sociocultural and biological influences on pain and pain-related responses. In subsequent studies, new participants ("perceivers") will view images of these initial participants ("targets") and will provide estimates of 'targets' pain experience. We will measure a) whether perceivers can accurately estimate 'targets' pain experience; b) whether accuracy differs as a function of similarity between target and perceiver (ingroup vs outgroup); and c) whether individuals can improve accuracy through feedback.

Outcome measures

Primary outcome measures for all experiments will be decisions about pain (experienced by self or other) measured with visual analogue scales, reaction time, and/or categorical judgments (pain/no pain). We will also measure physiological responses (e.g., facial muscle response, skin conductance, pupil dilation) and brain responses using functional magnetic resonance imaging (fMRI) as secondary outcome measures. We will test whether pain and pain-related responses varies as a function of sociocultural/demographic factors (e.g. race, ethnicity, sex) and whether accuracy in assessing others' pain is influenced by group similarity (i.e. ingroup vs. outgroup) and training (e.g. performance-related feedback)....

DETAILED DESCRIPTION:
Objective

The current proposal investigates behavioral, psychophysiological, and social processes that may help explain biases and disparate outcomes in pain. Health disparities, or health outcomes that adversely affect disadvantaged populations, are pervasive and apparent in many diseases and symptoms, including pain. Pain is the number one reason individuals seek medical treatment. Health disparities in pain encompass both differences in pain experience and treatment for pain. For instance, research indicates that Black individuals report increased pain and have reduced pain tolerance relative to White individuals, yet doctors are less likely to treat minority patients' pain and underestimate their pain experience. This project aims to address this systemic discrepancy by focusing on interpersonal processes that may contribute to these disparities, including socially-relevant responses to pain (i.e. pain expression) and pain assessment (e.g. visual attention). The proposed research aims to determine whether the study of pain expressions and their assessment can yield insights on how social factors shape pain and its treatment. Further, we test the efficacy of potential interventions designed to improve accuracy and reduce biases in pain assessment. If successful, this work will form the foundation of a new research program that will link the field of pain research with the field of social neuroscience, and forge new insights on the critical problem of health disparities in pain.

Study population

We will accrue up to 700 total healthy volunteers to target 240 completers.

Design

Our overall aim is to understand how social factors influence the assessment and management of pain, and to gain insight into psychosocial processes that may underlie health disparities in pain. We propose a series of studies designed to test these links. First, we will measure pain perception and physiological responses to painful stimuli in a diverse group of individuals to test for sociocultural and biological influences on pain and pain-related responses. In subsequent studies, new participants ("perceivers") will view images of these initial participants ("targets") and will provide estimates of 'targets' pain experience. We will measure a) whether perceivers can accurately estimate 'targets' pain experience; b) whether accuracy differs as a function of similarity between target and perceiver (ingroup vs outgroup); and c) whether individuals can improve accuracy through feedback.

Outcome measures

Primary outcome measures for all experiments will be decisions about pain (experienced by self or other) measured with visual analogue scales, reaction time, and/or categorical judgments (pain/no pain). We will also measure physiological responses (e.g., facial muscle response, skin conductance, pupil dilation) and brain responses using functional magnetic resonance imaging (fMRI) as secondary outcome measures. We will test whether pain and pain-related responses varies as a function of sociocultural/demographic factors (e.g. race, ethnicity, sex) and whether accuracy in assessing others' pain is influenced by group similarity (i.e. ingroup vs. outgroup) and training (e.g. performance-related feedback).

ELIGIBILITY:
* INCLUSION CRITERIA:

All Sub-Studies:

* Healthy
* Between 18 and 60 years old
* Fluent in English
* Able to provide written informed consent

EXCLUSION CRITERIA:

All Sub-Studies:

* Unable to comply with study procedures
* Has a major-medical condition or medical history that in a clinician's assessment could affect ability to comply with study procedures, including neurological conditions (including stroke, blindness or deafness, or a history of brain damage)
* Has a current mood disorder, anxiety disorder, or substance use disorder, or has a history of psychosis, hospitalization for a mental health condition, or recurrent psychiatric episodes.
* NIH staff member who is a subordinate/relative/co-worker of any investigator on the protocol
* Prior completion of a different sub-study within this protocol.
* Is born outside of the states or territories of the United States of America
* Does not currently reside in a state or territory of the United States of America

Sub-study 1:

* Has a major-medical condition or medical history that in a clinician's assessment could affect heat sensitivity or pain thresholds. This may include cardiovascular, autonomic, or neurological conditions or a chronic systemic disease (e.g., diabetes)
* Has a medical condition that in a clinician's assessment might affect somatosensation (e.g., Raynaud's disease, peripheral neuropathy, or circulatory disorder)
* Has a current chronic pain condition or has had chronic pain in the past (painful condition lasting more than six months)
* Has a dermatological condition affecting the testing region, such as scars, burns, or recent tattoos that might influence cutaneous sensibility
* Regular use of prescription medication that has a significant effect on pain or heat perception. Excluded medications include central-acting agents such as opiates (morphine, tramadol), antidepressants (amitriptyline, duloxetine, milnacipran), anticonvulsants (gabapentin, pregabalin), anxiolytics (barbituates, benzodiazepines), hypnotics (zolpidem, sodium oxybate), antipsychotics (valproate, lithium, olanzapine), antimigraine agents (sumatriptan, ergotamine), and muscle relaxants (cyclobenzaprine, carisoprodol). Use of analgesic medications, such as non-steroidal anti-inflammatories, salicylates, and acetaminophen, taken on an "as needed" basis is acceptable as long as the last dose was not taken was within 5 half-lives of testing.
* Is left handed

Sub-study 4, FMRI participants:

* Has a current chronic pain condition or has had chronic pain in the past (painful condition lasting more than six months)
* Is left-handed
* Any FMRI contraindications, including:

  * Ferromagnetic metal in the cranial cavity or eye, e.g. aneurysm clip, implanted neural stimulator, cochlear implant, ocular foreign body.
  * Implanted cardiac pacemaker or auto-defibrillator.
  * Insulin pump.
  * Irremovable body piercing.
* Pregnant women (based on urine test completed within 24 hours prior to scan).
* Those with an abnormality on a structural MRI that has functional consequences based on clinician assessment.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 700 (Estimated)
Dates: Start 2018-05-09 (Actual); Primary Completion 2027-05-17 (Estimated); Study Completion 2027-05-30 (Estimated)

PRIMARY OUTCOMES:
Physiological responses (facial muscle movement, skin conductance, respiration, pupil dilation, eye gaze position) | Every visit
  We measure facial responses to painful stimuli in substudy 1 and eye position in substudy 2 and 3.
Pain perception (pain ratings) | Every visit
  Individuals report their perceived pain or the pain they associate with other people they are viewing.

SECONDARY OUTCOMES:
Questionnaire measures (e.g. Fear of Pain questionnaire, McGill pain questionnaire) | Every visit
  We collect measures of identity and endorsement of beliefs about pain.

CONTACTS AND LOCATIONS:
Overall Officials: Lauren Y Atlas, Ph.D., Principal Investigator — National Center for Complementary and Integrative Health (NCCIH)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified data will be shared with other researchers as per the protocol. Identifiable data (i.e. images of faces) from participants who consent to data sharing may be shared with other researchers. Finally, identifiable data from participants who opt to be included in a stimulus set through the sub-study 1 consent form can be shown to other participants and in other studies to measure evaluation of facial responses to pain.
Supporting Information: ICF, CSR, Analytic Code
Time Frame: Face stimuli are available following completion for viewing by other study participants. Deidentified data will be made available upon publication.
Access Criteria: please see above.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2017-AT-0155.html